CLINICAL TRIAL: NCT02827227
Title: Values of the Immune Activation Markers CD38 and HLA-DR and the Ratio CD4/CD8 According to the Delay of Combined AntiRetroviral Therapy (c-ART) Initiation in Primary HIV-infected Patients (PRIMIMMUNO)
Acronym: PRIMIMMUNO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D21969
Record Dates: First submitted 2016-07-04; First posted 2016-07-11 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: HIV-infected Patients
Keywords: HIV-infected patients; cART; immune restoration; markers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary HIV- Infected patients: Primary HIV- Infected patients with a minimum of 2 years of effective cART.
  Interventions: Biological: lymphocytes immunophenotyping

INTERVENTIONS:
Biological: lymphocytes immunophenotyping — The lymphocytes immunophenotyping were performed from fresh EDTA-anticoagulated blood harvested during a routine follow-up of patients in HIV Lyon centers.
  HIV patients with a known history of PHI and a minimum of 2 years of effective cART (< 200 copies/mL) without interruption or virological failure were included in 2 centers in Lyon (Croix-Rousse and Edouard Herriot hospital).
  Baseline factors at the time of PHI, delay, type and duration of first and duration of total cART, CMV status, nadir CD4 cells count and level of activation markers on CD4 and CD8 cells (CD38 and HLA-DR) at the time of the study were assessed.
  Patients with hepatitis C or B virus co-infection or with a history of neoplasia or immunosuppressive therapy after the date of PIH were excluded.

SUMMARY:
The objective was to identify factors associated with the normalization of the CD4/CD8 ratio (>=1) in patients with a history of primary HIV infection (PHI) and long-term combined antiretroviral therapy (cART).

ELIGIBILITY:
Inclusion Criteria:

all HIV patients with a known history of PHI and a minimum of 2 years of effective cART (< 200 copies/mL) without interruption or virological failure

Exclusion Criteria:

Patients with hepatitis C or B virus co-infection or with a history of neoplasia or immunosuppressive therapy after the date of PIH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV patients
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2014-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
percentage of CD4+ and CD8+ T lymphocytes with activation markers (CD38 + and HLA-DR) | Day 0
  percentage of CD4+ and CD8+ T lymphocytes with activation markers (CD38 + and HLA-DR) according to the delay of cART initiation (early 3 months or delayed > 3 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon / Hôpital de la Croix Rousse, Lyon, France